CLINICAL TRIAL: NCT02405624
Title: Efficacy of Continuous Positive Airway Pressure of Treatment of Hypernasality of Children With Infantile Pompe Disease
Brief Title: CPAP for Infantile Pompe Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, MD, PhD, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201401043RINA
Record Dates: First submitted 2015-03-21; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP training (Experimental): Patients will be instructed and follow the continuous positive airway pressure (CPAP) training procedure
  Interventions: Procedure: continuous positive airway pressure

INTERVENTIONS:
Procedure: continuous positive airway pressure — CPAP training for muscle strength

SUMMARY:
Patients with infantile onset Pompe disease will be trained with continuous positive airway pressure to see if hypernasality can be improved.

ELIGIBILITY:
Inclusion Criteria:

1. confirm as Pompe disease
2. Age 4 and can speak 2-words sentence by order
3. mild to severe hypernasality
4. have regular speech therapy for 8 weeks or longer

Exclusion Criteria:

(1）hearing loss （2）congenital pharyngeal or laryngeal structure anomalies including cleft palate （3）cerebral palsy （4）recent otitis media effusion （5）very severe hypernasality （6）use non-invasive ventilator

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
decrease in hypernasality | 6 months
  score hypernasality degree and compare

SECONDARY OUTCOMES:
increase in speech intelligibility | 6 months
  score speech intelligibility degree and compare

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan